CLINICAL TRIAL: NCT03572205
Title: Fatty Acid Desaturase Gene Locus Interactions With Diet (FADSDIET2)
Acronym: FADSDIET2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FADSDIET2
Record Dates: First submitted 2018-06-13; First posted 2018-06-28 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Fatty Acids; Genetics
Keywords: Nutrigenetics
MeSH Terms: interventions — Sunflower Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CC genotype LA (Experimental): 4-week study diet will be isocaloric following the habitual diet of the participants with a supplement of 30-50 ml (5-6 % of energy intake) of sunflower oil (source of LA: linoleic acid) daily, depending on body weight. The same diet will be instructed for both genotypes.
  Interventions: Dietary Supplement: LA
- TT genotype LA (Experimental): 4-week study diet will be isocaloric following the habitual diet of the participants with a supplement of 30-50 ml (5-6 % of energy intake) of sunflower oil (source of LA: linoleic acid) daily, depending on body weight. The same diet will be instructed for both genotypes.
  Interventions: Dietary Supplement: LA
- CC genotype ALA (Experimental): 4-week study diet will be isocaloric following the habitual diet of the participants with a supplement of 30-50 ml (5-6 % of energy intake) of camelina oil (source of alpha-linolenic acid: ALA) daily, depending on body weight. The same diet will be instructed for both genotypes.
  Interventions: Dietary Supplement: ALA
- TT genotype ALA (Experimental): 4-week study diet will be isocaloric following the habitual diet of the participants with a supplement of 30-50 ml (5-6 % of energy intake) of camelina oil (source of alpha-linolenic acid: ALA) daily, depending on body weight. The same diet will be instructed for both genotypes.
  Interventions: Dietary Supplement: ALA

INTERVENTIONS:
Dietary Supplement: LA — The source of linoleic acid (LA) will be sunflower oil (62-63 % LA). The study diets will be isocaloric. The allowed weight change during the study is ± 2-3 %. The amount of supplementary oil will be calculated individually based on the calculated energy expenditure and adjusted, if necessary, during the study based on body weight measurements.
  Other Names: sunflower oil
  Arms: CC genotype LA; TT genotype LA
Dietary Supplement: ALA — The source of alpha-linolenic acid (ALA) will be camelina sativa oil (30-35 % ALA). The study diets will be isocaloric. The allowed weight change during the study is ± 2-3 %. The amount of supplementary oil will be calculated individually based on the calculated energy expenditure and adjusted, if necessary, during the study based on body weight measurements.
  Other Names: camelina oil
  Arms: CC genotype ALA; TT genotype ALA

SUMMARY:
Interactions between genes and environment, are likely to be crucial in the development of the common diseases such as type 2 diabetes. Recently, the investigators have obtained data that genotypes of genes encoding for fatty acid desaturases 1 and 2 (FADS1 and FADS2) are the strongest genes in a genome-wide analysis regulating serum fatty acid profile.The aim of this study is to test if subjects with different genotypes of the FADS2 gene respond differently to a diet supplemented with linoleic acid or alpha-linolenic acid (substrates for FADS2). The study hypothesizes that subjects will be more sensitive to the dietary modifications according to their genotype leading to more robust differences in serum FA profile, tissue inflammation and serum lipids.

DETAILED DESCRIPTION:
Lean and overweight subjects (Body mass index: BMI >20kg/m2 <32kg/m2 ) with CC and TT genotypes of FADS1 single nucleotide polymorphism (SNP) from the METabolic Syndrome in Men (METSIM) study, in which currently >10000 men are included from the population living in Kuopio, will be recruited. Seventy subjects with CC genotype will be selected after matching with the 70 subjects with the TT genotype for age and BMI.

After a 4-week run-in period, the subjects within each genotype group will be randomly assigned into two study groups according to medians of BMI, age and fasting plasma glucose concentration: in one group the diet will be enriched with linoleic acid (LA, sunflower oil) and in the other group with alpha-linolenic acid (ALA, camelina oil). The intervention will last for 8 weeks.

The sample size calculation is based on the observed change in arachidonic acid (AA) in the cholesterol esthers fraction between CC and TT genotypes (12.14 vs. 4.20 mol%, respectively) after the diet enriched in LA from preliminary data. Considering a β=0.80 and an α=0.025 instead of only 0.05 to account for the fact that we now have two dietary interventions instead of one, 31 participants in each study group would need to be included. Assuming around 15% of dropouts in this trial, a final sample size of 35 for each group is required.

The study diet will be isocaloric following the habitual diet of the participants with a supplement of 30-50 ml (25-45 g) sunflower or camelina oil daily depending on body weight. The dose of each oil is not known to cause any side effects or adverse events and even higher doses have been safe.

Participants will record their daily oil consumption and 4-day food records will be collected at the beginning and two times during the intervention period to measure daily intake of macronutrients and specifically different fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Participants of METSIM study cohort with CC/TT FADS1 rs174547 SNP genotype.
* BMI 20-32 kg/m2.
* Healthy .

Exclusion Criteria:

* Diagnosis of type 2 diabetes.
* Diagnosis of chronic diseases and conditions, that may hamper the ability to follow the dietary intervention protocol
* Chronic liver, thyroid and kidney diseases
* Alcohol abuse (> 40 g/d)
* BMI >32 kg/m2.

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men because the population source for recruitment Metabolic syndrome in men (METSIM) study is composed solely by men.
Enrollment: 140 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Change in fatty acid composition of serum lipid fractions | 8 weeks
  Fatty acid composition of serum lipid fractions

SECONDARY OUTCOMES:
Glucose and insulin metabolism response | 8 weeks
  Oral glucose tolerance test (OGTT) variables: fasting, 30 min and 120 min glucose and insulin measurements
Inflammatory markers response | 8 weeks
  Serum circulating levels of high-sensitivity C-reactive protein
Adipose tissue biopsies | 8 weeks
  Subcutaneous adipose tissue taken by open biopsy to collect 1-5 g of adipose tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Pihlajamäki, MD, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No